CLINICAL TRIAL: NCT04291963
Title: De-epithelialized Gingival Graft Versus Subepithelial Connective Tissue Graft in the Treatment of Multiple Adjacent Gingival Recessions Using the Tunnel Technique
Brief Title: The Efficacy of De-epithelialized Free Gingival Graft on Treatment of Multiple Gingival Recessions With Tunnel Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sıla Çağrı İşler, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36290600/110
Record Dates: First submitted 2020-02-24; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Gingival Recession
Keywords: gingival recessions; connective tissue graft; de-epithelialized gingival graft; tunnel technique
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DGG + TUN (Active Comparator): The multiple adjacent gingival recession sites were treated with DGG in conjunction with TUN technique.
  Interventions: Procedure: DGG + TUN
- SCTG + TUN (Active Comparator): The multiple adjacent gingival recession sites were treated with SCTG in conjunction with TUN technique.
  Interventions: Procedure: SCTG + TUN

INTERVENTIONS:
Procedure: DGG + TUN — In the DGG group, CTG was obtained at palatal mucosa by means of intra-oral de-epithelialization of the FGG using a 2.3 mm diameter diamond burr (801G/023, EMS, Aldrich Co., USA) with NaCL 0.9% saline irrigation
  Arms: DGG + TUN
Procedure: SCTG + TUN — In SCTG group, graft was harvested through the single-incision approach at palatal mucosa
  Arms: SCTG + TUN

SUMMARY:
The predictable treatment of multiple adjacent gingival recessions (MAGRs) represents a major challenge in periodontal plastic surgeries due to MAGRs' complicated predisposing anatomic features, such as thin gingival phenotype or limited keratinized tissue. The present study aimed to investigate the clinical efficacy and postoperative morbidity of de-epithelialized gingival graft (DGG) compared to subepithelial connective tissue graft (SCTG) on the treatment of multiple adjacent gingival recessions (MAGRs) with tunnel technique (TUN). A total of 38 patients, who have been referred to the Gazi University Faculty of Dentistry Department of Periodontology, were randomly assigned to receive TUN in combination with either DGG or SCTG. Clinical measurements were recorded at baseline and at 3, 6 and 12 months after surgeries. Immediately after surgery, a questionnaire was given to each patient evaluating postoperative pain, patients' discomfort, sensitivity and bleeding at 1, 2, 3, 7, 14 and 28 days after surgery. Moreover, the characteristics of the grafts harvested by these two different techniques were evaluated histopathologically and histomorphometrically.

DETAILED DESCRIPTION:
The predictable treatment of multiple adjacent gingival recessions (MAGRs) represents a major challenge in periodontal plastic surgeries due to MAGRs' complicated predisposing anatomic features, such as thin gingival phenotype or limited keratinized tissue, variations in the depth and width of the adjacent recession defects, shallow vestibules and high frenum attachments. Furthermore, in these cases, wound healing is often more difficult due to factors such as larger avascular surface and poor blood supply.

The coronally advanced flap (CAF) or the tunnel technique (TUN) with graft-based subepithelial connective tissue procedures have been reported to be the most predictable methods for the treatment of MAGRs. On account of the advantages of TUN, including superior blood supply and advanced wound healing owing to its conservative characteristics associated with the flap elevation without papillae dissection or vertical releasing incisions, this approach has recently achieved popularity compared to other methods.

Although the use of connective tissue grafts (CTGs), together with various surgical techniques, has been accepted as "the gold standart" for the treatment of GRs, some disadvantages of CTG are underlined. Limited donor tissue in the cases where inadequate amount of palatal tissue thickness and/or a bigger dimension of CTG is needed, as in the treatment of MAGRs are claimed to be among those disadvantages (Zucchelli et al., 2010). Moreover, subepitelial CTG (SCTG), either harvested by 'trap-door' (TD) or 'single-incision' (SI) approaches, have been frequently associated with post-operative pain and discomfort, as well as palatal flap necrosis/dehiscence at the donor site.

To overcome these limitations, and obtain a firmer and uniform CTG, de-epithelializing of the free gingival grafts (FGG) have been proposed, especially when palatal fibromucosal tissue thickness is inadequate (≤2.5 mm) and a large graft dimension in apico-coronal or mesio-distal directions is required. De-epithelialized gingival graft (DGG) have also been suggested to have less prone to post-operative shrinkage, because of obtaining larger amount of collagen-rich connective tissue from lamina propria, minimal amount of fatty/glandular tissue and less number of medium to large vessels. Previously it was reported that DGG applied with the TUN presented better manuplation in recipent area and reduced postoperative morbidity compared to a conventional CTG, and resulted in a successful root coverage outcome with increased both width and thickness of the keratinized tissue in the treatment of MAGRs. In a randomized clinical trial (RCT), Zuchelli et al. found no significant differences regarding post-operative pain and root coverage outcomes when compared SCTG and DGG in combination with CAF in the treatment of single or multiple GRs. However, a significant difference was observed in terms of keratinized tissue thickness (KTT) in favor of DGG, and this finding was attributed to the its characteristics of better stability, low shrinkage rates and to allow the incorporation of the portion of connective tissue closest to the epithelium. Despite all biologically advantages of DGG, there is scarce information in the literature on its clinical significance in combination with TUN compared to conventional CTG procedures in the treatment of MAGRs. Therefore, the present study aimed to investigate the clinical efficacy and postoperative morbidity of DGG compared to SCTG on treatment of MAGRs with TUN. The primary objective was to assess the root coverage outcomes of DGG versus SCTG with TUN at 1-year postoperatively. The secondary objectives were to evaluate postoperative patient morbidity of these procedures and the characteristics of the grafts harvested by these two different techniques histopathologically and histomorphometrically.

ELIGIBILITY:
Inclusion Criteria:

* • Age between 18 - 60 years,

  * Non-smoker and systemically healthy,
  * No active periodontal disease,
  * Presence of at least two single-rooted teeth with Miller class I and/or II (RT1) (Cairo, Nieri, Cincinelli, Mervelt, & Pagliaro, 2011; Miller, 1985) buccal gingival recession defects ≥2 mm in depth
  * Full mouth plaque and bleeding score of <15% and no probing depths >3 mm,
  * Absence of non-carious cervical lesions (NCCLs) and non-detectable cemento-enamel junction (CEJ) at the defect sites,
  * No history of previous periodontal plastic surgery at the affected sites.

Exclusion Criteria:

* • Presence of caries lesions or restorations in the cervical area,

  * Intake of medications which impede periodontal tissue health and healing,
  * Medical contraindications for periodontal surgical procedures,
  * Pregnancy and lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-12-09 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Root coverage outcomes | 1-year postoperatively
  Mean root coverage of DGG versus SCTG with TUN

SECONDARY OUTCOMES:
Root coverage outcomes | 1-year postoperatively
  Complete root coverage of DGG versus SCTG with TUN
Root coverage outcomes | 1-year postoperatively
  Recession depth
patient morbidity | up to 28 days postoperatively
  postoperative pain
patient morbidity | up to 28 days postoperatively
  patients' discomfort
histopathological features of the graft | through study completion, an average of 1 year
  graft cellularity
histopathological features of the graft | through study completion, an average of 1 year
  vascularization

CONTACTS AND LOCATIONS:
Overall Officials: Burcu C Ozdemir, Assoc Prof, Study Director — Gazi University
Locations (1):
- Sila Isler, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aroca S, Barbieri A, Clementini M, Renouard F, de Sanctis M. Treatment of class III multiple gingival recessions: Prognostic factors for achieving a complete root coverage. J Clin Periodontol. 2018 Jul;45(7):861-868. doi: 10.1111/jcpe.12923. Epub 2018 Jun 15. PMID 29757468
- [Result] Sculean A, Cosgarea R, Stahli A, Katsaros C, Arweiler NB, Miron RJ, Deppe H. Treatment of multiple adjacent maxillary Miller Class I, II, and III gingival recessions with the modified coronally advanced tunnel, enamel matrix derivative, and subepithelial connective tissue graft: A report of 12 cases. Quintessence Int. 2016;47(8):653-9. doi: 10.3290/j.qi.a36562. PMID 27446995
- [Result] Tatakis DN, Chambrone L, Allen EP, Langer B, McGuire MK, Richardson CR, Zabalegui I, Zadeh HH. Periodontal soft tissue root coverage procedures: a consensus report from the AAP Regeneration Workshop. J Periodontol. 2015 Feb;86(2 Suppl):S52-5. doi: 10.1902/jop.2015.140376. Epub 2014 Oct 15. PMID 25315018
- [Result] Tavelli L, Barootchi S, Nguyen TVN, Tattan M, Ravida A, Wang HL. Efficacy of tunnel technique in the treatment of localized and multiple gingival recessions: A systematic review and meta-analysis. J Periodontol. 2018 Sep;89(9):1075-1090. doi: 10.1002/JPER.18-0066. Epub 2018 Aug 13. PMID 29761502
- [Result] Aroca S, Molnar B, Windisch P, Gera I, Salvi GE, Nikolidakis D, Sculean A. Treatment of multiple adjacent Miller class I and II gingival recessions with a Modified Coronally Advanced Tunnel (MCAT) technique and a collagen matrix or palatal connective tissue graft: a randomized, controlled clinical trial. J Clin Periodontol. 2013 Jul;40(7):713-20. doi: 10.1111/jcpe.12112. Epub 2013 Apr 30. PMID 23627374
- [Result] Chambrone L, Tatakis DN. Periodontal soft tissue root coverage procedures: a systematic review from the AAP Regeneration Workshop. J Periodontol. 2015 Feb;86(2 Suppl):S8-51. doi: 10.1902/jop.2015.130674. PMID 25644302
- [Result] Buti J, Baccini M, Nieri M, La Marca M, Pini-Prato GP. Bayesian network meta-analysis of root coverage procedures: ranking efficacy and identification of best treatment. J Clin Periodontol. 2013 Apr;40(4):372-86. doi: 10.1111/jcpe.12028. Epub 2013 Jan 24. PMID 23346965
- [Result] Zucchelli G, Mele M, Stefanini M, Mazzotti C, Marzadori M, Montebugnoli L, de Sanctis M. Patient morbidity and root coverage outcome after subepithelial connective tissue and de-epithelialized grafts: a comparative randomized-controlled clinical trial. J Clin Periodontol. 2010 Aug 1;37(8):728-38. doi: 10.1111/j.1600-051X.2010.01550.x. Epub 2010 Jun 24. PMID 20590963
- [Result] Harris RJ. A comparison of two techniques for obtaining a connective tissue graft from the palate. Int J Periodontics Restorative Dent. 1997 Jun;17(3):260-71. PMID 9497718
- [Result] Bruno JF. Connective tissue graft technique assuring wide root coverage. Int J Periodontics Restorative Dent. 1994 Apr;14(2):126-37. PMID 7928129
- [Result] Hurzeler MB, Weng D. A single-incision technique to harvest subepithelial connective tissue grafts from the palate. Int J Periodontics Restorative Dent. 1999 Jun;19(3):279-87. PMID 10635174
- [Result] Lorenzana ER, Allen EP. The single-incision palatal harvest technique: a strategy for esthetics and patient comfort. Int J Periodontics Restorative Dent. 2000 Jun;20(3):297-305. PMID 11203571
- [Result] Griffin TJ, Cheung WS, Zavras AI, Damoulis PD. Postoperative complications following gingival augmentation procedures. J Periodontol. 2006 Dec;77(12):2070-9. doi: 10.1902/jop.2006.050296. PMID 17209793
- [Result] Gobbato L, Nart J, Bressan E, Mazzocco F, Paniz G, Lops D. Patient morbidity and root coverage outcomes after the application of a subepithelial connective tissue graft in combination with a coronally advanced flap or via a tunneling technique: a randomized controlled clinical trial. Clin Oral Investig. 2016 Nov;20(8):2191-2202. doi: 10.1007/s00784-016-1721-7. Epub 2016 Jan 27. PMID 26814715
- [Result] Isler SC, Eraydin N, Akkale H, Ozdemir B. Oral flurbiprofen spray for mucosal graft harvesting at the palatal area: A randomized placebo-controlled study. J Periodontol. 2018 Oct;89(10):1174-1183. doi: 10.1002/JPER.17-0381. Epub 2018 Aug 29. PMID 30007054
- [Result] Harris RJ. Root coverage in molar recession: report of 50 consecutive cases treated with subepithelial connective tissue grafts. J Periodontol. 2003 May;74(5):703-8. doi: 10.1902/jop.2003.74.5.703. PMID 12816304
- [Result] Bosco AF, Bosco JM. An alternative technique to the harvesting of a connective tissue graft from a thin palate: enhanced wound healing. Int J Periodontics Restorative Dent. 2007 Apr;27(2):133-9. PMID 17514885
- [Result] de Sanctis M, Baldini N, Goracci C, Zucchelli G. Coronally advanced flap associated with a connective tissue graft for the treatment of multiple recession defects in mandibular posterior teeth. Int J Periodontics Restorative Dent. 2011 Nov-Dec;31(6):623-30. PMID 22140664
- [Result] Zuhr O, Baumer D, Hurzeler M. The addition of soft tissue replacement grafts in plastic periodontal and implant surgery: critical elements in design and execution. J Clin Periodontol. 2014 Apr;41 Suppl 15:S123-42. doi: 10.1111/jcpe.12185. PMID 24640997
- [Result] Azar EL, Rojas MA, Patricia M, Carranza N. Histologic and Histomorphometric Analyses of De-epithelialized Free Gingival Graft in Humans. Int J Periodontics Restorative Dent. 2019 Mar/Apr;39(2):221-226. doi: 10.11607/prd.3544. PMID 30794258
- [Result] Bertl K, Pifl M, Hirtler L, Rendl B, Nurnberger S, Stavropoulos A, Ulm C. Relative Composition of Fibrous Connective and Fatty/Glandular Tissue in Connective Tissue Grafts Depends on the Harvesting Technique but not the Donor Site of the Hard Palate. J Periodontol. 2015 Dec;86(12):1331-9. doi: 10.1902/jop.2015.150346. Epub 2015 Aug 20. PMID 26291293
- [Result] Tavelli L, Barootchi S, Namazi SS, Chan HL, Brzezinski D, Danciu T, Wang HL. The influence of palatal harvesting technique on the donor site vascular injury: A split-mouth comparative cadaver study. J Periodontol. 2020 Jan;91(1):83-92. doi: 10.1002/JPER.19-0073. Epub 2019 Aug 18. PMID 31376154
- [Result] McLeod DE, Reyes E, Branch-Mays G. Treatment of multiple areas of gingival recession using a simple harvesting technique for autogenous connective tissue graft. J Periodontol. 2009 Oct;80(10):1680-7. doi: 10.1902/jop.2009.090187. PMID 19792859